CLINICAL TRIAL: NCT04684966
Title: Interest of Adding Neuromuscular Electrical Stimulation for Quadriceps Femoris and Triceps Surae Muscles to Pulmonary Rehabilitation in COPD : Randomized Clinical Trial
Brief Title: Combined Neuromuscular Electrical Stimulation for Quadriceps and Triceps During Pulmonary Rehabilitation in COPD
Acronym: COMBIELEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 29BRC20.0249
Record Dates: First submitted 2020-12-10; First posted 2020-12-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease Overlap Syndrome; Asthma
Keywords: Pulmonary Rehabilitation; Neuromuscular Electrical Stimulation; COPD; Muscular Strengthening
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (EG) (Experimental): Randomized intervention in the NMES (GE) group:
  Patients in the NMES group will receive, in addition to conventional rehabilitation, combined quadriceps femoris and triceps surae NMES.
  Detail of the NMES :
  * Stimulation is performed in a semi-seated position, biphasic current, 8 channels in total (possibility of 16 electrodes).
  * One device per lower limb of each patient is necessary: 4 electrodes are placed on the quadriceps and 4 electrodes on the triceps, on each lower limb.
  * Stimulation frequency: 50hz.
  * Pulse duration: 400 μs.
  * Contraction time: 6 seconds.
  * Rest time: 6 seconds.
  * The intensity must generate a visible muscular contraction and must be well supported. by the patient.
  * The voluntary contraction accompanies the electrical stimulation.
  * Surface electrode 50 × 50 mm.
  Interventions: Device: Neuromuscular Electrical Stimulation
- Control group (CG) (Sham Comparator): Patients in the control group (GC) will receive, in addition to the classical rehabilitation, the combined sham NMES of the quadriceps femoris and triceps surae.
  Detail of the NMES :
  * It is carried out 5 times a week for 4 weeks, supervised by a physiotherapist.
  * The device used will be the same as in the EG group.
  * Stimulation is performed in a semi-seated position, biphasic current, 8 channels in total (16 electrodes can be used).
  * One device per lower limb of each patient is required: 4 electrodes are placed on the quadriceps and 4 electrodes on the triceps, on each lower limb.
  * Stimulation frequency: 5hz.
  * Pulse duration: 100 μs.
  * Contraction time: 6 seconds.
  * Rest time: 6 seconds.
  * The intensity must generate a visible muscle contraction and must be well supported by the patient.
  * The voluntary contraction accompanies the electrical stimulation.
  * Surface electrode 50 × 50 mm.
  Interventions: Device: Sham Neuromuscular Electrical Stimulation

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Standart pulmonary rehabilitation with combined quadriceps and triceps surae ESNM using two identical electrotherapy devices allowing simultaneous stimulation of the quadriceps and triceps (EG group).
  Arms: Experimental group (EG)
Device: Sham Neuromuscular Electrical Stimulation — Standart pulmonary rehabilitation with combined sham NMES of the quadriceps and triceps surae performed using two identical electrotherapy devices allowing simultaneous stimulation of the quadriceps and triceps (CG group)
  Arms: Control group (CG)

SUMMARY:
Patients with COPD frequently have muscle disorders. Pathogenic mechanisms generate significant pathophysiological changes in the locomotor muscles structure, leading to decreased strength, decreased endurance and limited exercise capacity.

Pulmonary rehabilitation is the first choice therapy and training overall lower limb endurance is a priority. Even if the effects of pulmonary rehabilitation are no longer to be demonstrated, it is still necessary to optimize the modalities of muscular strengthening. In fact, it is recommended to associate to this global endurance training a specific strengthening of the muscles of the lower limbs. Neuromuscular electrostimulation (NMES) is a muscular strengthening technique, but this method is not used in usual practice in pulmonary rehabilitation and often only the quadriceps are concerned. In a pulmonary rehabilitation program, including sessions of NMES of the quadriceps femoris and triceps surae could increase its effectiveness.

Recent studies suggest that NMES can improve muscle function, exercise tolerance, dyspnea and quality of life in COPD patients.

A pilot study compared the effects of the combined quadriceps femoris and triceps surae versus quadriceps alone. The final evaluation showed a greater improvement in exercise capacity in favour of the combined NMES group. Only two studies with small numbers of patients evaluated the effect of combined quadriceps femoris and triceps surae NMES in pulmonary rehabilitation, with encouraging results in terms of functional gain. Further larger studies seem necessary to evaluate the effects of combined quadriceps femoris and triceps surae NMES in pulmonary rehabilitation. The objective of the study is to show that combined quadriceps femoris and triceps surae NMES during a pulmonary rehabilitation program provides a more significant improvement in exercise capacity compared to a standard pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD stages 2 to 4 (A to D) admitted to the Pulmonary Rehabilitation Department of the "Centre Hospitalier des Pays de Morlaix" or the "CHRU of Brest".
* Patient aged 18 years or older.
* Patient able to consent and having signed a consent form.

Exclusion Criteria:

* Patient with a history of pneumonectomy, lobectomy dated less than 6 months old
* Patient with an inability to complete a respiratory rehabilitation program in its entirety
* Patient under guardianship or curatorship
* Person equipped with electronic devices such as pacemakers and intracardiac defibrillators.
* Skin lesions and infectious foci on the area where the electrodes.
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Walking distance change | Day 0 and Day 28
  Assessment of the walking distance (in meters) covered during the 6-minute walking test before and after rehabilitation (between D0 and D28± 4 days). The main endpoint is the change (in meters) between Day 0 and Day 28.

SECONDARY OUTCOMES:
Maximal isometric voluntary quadriceps strengh | Day 0 and Day 28
  Maximal isometric voluntary quadriceps strengh assessment (in newton) with handheld dynamometer
Maximal isometric voluntary endurance change | Day 0 and Day 28
  Maximal isometric voluntary endurance assessment with handheld dynamometer
Maximal isometric voluntary triceps surae strengh change | Day 0 and Day 28
  Maximal isometric voluntary triceps surae strengh assessment (in newton) with dynamometer type MICROFET 2 before and after rehabilitation.
Exercise capacity change with the 1 min sit to stand test | Day 0 and Day 28
  Exercise capacity assessment during the 1 min sit to stand test before and after rehabilitation.
Exercise capacity change with the 6 min step test | Day 0 and Day 28
  Exercise capacity assessment during the 6 min step test before and after rehabilitation.
Exercise capacity change with the incremental shuttle test | Day 0 and Day 28
  Exercise capacity assessment during the incremental shuttle test before and after rehabilitation.
Exercise capacity change with the endurance shuttle walk test | Day 0 and Day 28
  Exercise capacity assessment during the endurance shuttle walk test before and after rehabilitation.
  before and after rehabilitation.
Dyspnea change during the 6-minute walking test | Day 0 and Day 28
  Dyspnea assessment at the end of the 6-minute walking test, with the Borg scale, before and after rehabilitation
Dyspnea change during the 6-minute walking test | Day 0 and Day 28
  Dyspnea assessment at the end of the 6-minute walking test, with the Multidimensional dyspnea profile questionnaire, before and after rehabilitation
Isotime dyspnea change with the endurance shuttle walk test | Day 28
  Isotime dyspnea assessment during the endurance shuttle walk test, using Borg scale after rehabilitation.
Dyspnea change with the mMRC (modified Medical Research Council) scale | Day 0 and Day 28
  Assessment of dyspnea with the mMRC scale (min : 0 ; max : 4), before and after rehabilitation.
Dyspnea change with the LCADL (London Chest Activity of Daily Living) questionnaire | Day 0 and Day 28
  Assessment of dyspnea with the LCADL questionnaire (better score : 0; worse score: 5), before and after rehabilitation.
Dyspnea change with the Dyspnea-12 questionnaire | Day 0 and Day 28
  Assessment of dyspnea with the Dyspnea-12 questionnaire, before and after rehabilitation.
Quality of life change with the St George's Respiratory Questionnaire | Day 0 and Day 28
  Quality of life assessment with the St George's Respiratory Questionnaire, before and after rehabilitation.
Quality of life change with the CAT (COPD Assessment Test) Questionnaire | Day 0 and Day 28
  Quality of life assessment with COPD Assessment Test (better : 0; worse : 5), before and after rehabilitation.
Fear of fall change with the FES (Falls Efficacy Scale) questionnaire | Day 0 and Day 28
  Fear of fall (FES-I Questionnaire) assessment (better : 1; worse : 4), before and after rehabilitation.
Anxiety disorder change | Day 0 and Day 28
  Anxiety disorder assessment (HAD questionnaire) (better : 0; worse : 3) before and after rehabilitation.
Depressive disorder change | Day 0 and Day 28
  Depressive disorder assessment (HAD questionnaire) (better : 0; worse : 3) before and after rehabilitation.
Non fat mass index change | Day 0 and Day 28
  Assessment of the non fat mass index with impedancemetry , before and after rehabilitation.
Self esteem change | Day 0 and Day 28
  Self esteem assessment with PSI-6 (Physical Self Inventory) questionnaire (worse :0 ; better :10)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU La Cavale Blanche, Brest, France, France

IPD SHARING:
Plan to Share IPD: Undecided